CLINICAL TRIAL: NCT01342380
Title: Pharmacogenetic Study of Pioglitazone and Quetiapine XR Treatment Response in Mood Disorders
Brief Title: Pioglitazone and Quetiapine XR Pharmacogenetic Study
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: #10-10-25
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Bipolar Disorder; Major Depressive Disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Seroquel: Participants who received Seroquel
- Pioglitazone: Participants who received pioglitazone

SUMMARY:
Obtain phenotypic data and a DNA/blood sample from mood disorder patients undergoing pioglitazone or quetiapine XR treatment as a part of an IRB approved clinical trial conducted at the Mood Disorders Program. Pioglitazone treatment is examined in metabolic syndrome comorbid with bipolar depression (IRB # 07-08-24) and unipolar depression (IRB # 07-07-20). Quetiapine XR treatment is examined in generalized anxiety disorder comorbid with bipolar depression (IRB # 10-06-19) and unipolar depression (IRB # 12-01-29). Please refer to the respective IRB protocols for more information.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated in IRB protocols 10-06-19, 12-07-29, 07-07-20, and 07-08-24
* Patient must give consent to participate, sign and date the IRB approved written informed consent form prior to the initiation of any procedures for this study
* Patient must be diagnosed with Bipolar Disorder or Major Depressive Disorder
* Patient must be at least 18 years old
* Patient must be willing to give a blood sample

Exclusion Criteria:

* Patient lacks the capacity to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 310 subjects between the ages of 18 and 70 will be targeted for enrollment. We anticipate a low enrollment rate of 200 from the targeted 310 participants. Eligible participants will be diagnosed with DSM-IV bipolar disorder (type I, II, or not otherwise specified) or DSM-IV major depressive disorder, as determined by extensive clinical interview and the Mini-International Neuropsychiatric Interview-Plus (MINI-Plus). Participants will be approached for enrollment if they are currently enrolled in one of four studies: IRB protocol numbers 10-06-19, 12-07-29, 07-07-20, and 07-08-24. Please see these protocols for additional study specific information.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2011-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Genetic markers associated with treatment response | Up to 1.5 years
  Genetic markers in PPARG, 5-HT2A, CYP3A4 and CYP2C8 genes known to be related in the pharmacodynamics and pharmacokinetics of pioglitazone or quetiapine XR will be associated with treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Fan, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States